CLINICAL TRIAL: NCT04668157
Title: A Phase 3, Open-label, Multicenter, Long-term Study to Evaluate the Safety, Efficacy and Pharmacokinetics of TAK-536 in Pediatric Subjects From 2 to Less Than 6 Years of Age With Hypertension
Brief Title: A Study of TAK-536 in Children From 2 to Less Than 6 Years Old With High Blood Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Azilsartan-3004; U1111-1259-9316 (Other: WHO); jRCT2041200083 (Registry Identifier: jRCT)
Record Dates: First submitted 2020-12-10; First posted 2020-12-16 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — azilsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAK-536 (Experimental): TAK-536 granule formulation, orally once daily before or after breakfast. The initial dose of TAK-536 will be 0.1 mg/kg (not exceeding 2.5 mg/day). After the initial dose, TAK-536 will be titrated to 0.2 mg/kg (not exceeding 5 mg/day), 0.4 mg/kg (not exceeding 10 mg/day), and 0.8 mg/kg (not exceeding 20 mg/day) if the subjects do not achieve the target blood pressure and no concerns are found in safety and tolerability.
  Interventions: Drug: TAK-536

INTERVENTIONS:
Drug: TAK-536 — TAK-536 granule formulation

SUMMARY:
The main aim of this study is to check the safety of TAK-536. This study will take place in Japan. At the first visit, the study doctor will check if each child can take part. For those who can take part, each participant will have a check-up by the study doctor. After this, each participant will take placebo. This might take 2 weeks.

After this, parents or the caregivers of each participant will be given sachets that contain granules of TAK-536 to give to that participant. The participants will take the TAK-536 granules once a day for 52 weeks.

After treatment has finished, participants will visit the study clinic for a final check-up.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-536. TAK-536 is being tested in pediatric participants with hypertension aged 2 to less than 6 years. This study will look at the safety, efficacy, and pharmacokinetics of long-term administration of TAK-536.

The study will enroll 10 participants. Participants will receive the study drug (TAK-536) orally once daily before or after breakfast.

The initial dose of TAK-536 will be 0.1 mg/kg (not exceeding 2.5 mg/day). After the initial dose, TAK-536 will be titrated to 0.2 mg/kg (not exceeding 5 mg/day), 0.4 mg/kg (not exceeding 10 mg/day), and 0.8 mg/kg (not exceeding 20 mg/day) if the participants do not achieve the target blood pressure and no concerns are found in safety and tolerability.

This multi-center trial will be conducted in Japan. The overall time to participate in this study is approximately 56 weeks. Participants will make multiple visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator or subinvestigator, the participant's parent or legal guardian is capable of understanding and complying with protocol requirements.
2. The participant's parent or the participant's legal guardian is capable of signing and dating a written informed consent form on behalf of the participant prior to the initiation of any study procedures.
3. A Japanese participant who has a diagnosis of hypertension. A participant is eligible if he/she is deemed hypertensive according to the reference blood pressure values of children by gender and age; office sitting diastolic or systolic blood pressure >=95th percentile for essential hypertension without concomitant hypertensive organ damage, and >=90th percentile for secondary hypertension with concomitant CKD, diabetes mellitus, heart failure or hypertensive organ damage.

   In addition, participants need to meet the following criteria:

   If currently treated with any antihypertensive drugs at the start of the Run-in Period: Participant has a documented diagnosis of hypertension and an office sitting diastolic or systolic blood pressure meeting the above criteria at the end of the Run-in Period (Week 0).

   If currently untreated with any antihypertensive drugs at the start of the Run-in Period: Participant meets the above criteria for hypertension on 3 separate time points including screening and the end of the Run-in Period (Week 0). In addition, for a participant with essential hypertension without hypertensive organ damage, the participant does not respond to non-pharmacological therapy such as diet modification or exercises for at least 3 months within 1 year prior to the start of screening.
4. The participant is male or female and aged 2 to less than 6 years at the time of informed consent.
5. At screening, the participant has not less than minus 2 standard deviations from mean weight for age of reference population shown in the table of pediatric body weight by the Japanese Society for Pediatric Endocrinology.
6. The participant is able to swallow the study drug.
7. A participant who has undergone kidney transplantation is eligible if he/she underwent the transplantation, and the graft has been functionally stable (estimated glomerular filtration rate [eGFR] >= 30 mL/min/1.73 m^2) for at least 6 months with evidence (eg, Doppler echography, CT [computed tomography] scan or MRI [magnetic resonance imaging]) excluding dose at least 30 days prior to screening is eligible.
8. The participant, judged by the investigator or subinvestigator, who can safely discontinue the therapy with RAS inhibitors for 2 weeks prior to the Treatment Period. This period may change to between 1 and 4 weeks depending on the participant's duration of Run-in Period.

Exclusion Criteria:

1. The participant has received any investigational compound within 30 days prior to screening or is participating in another clinical study or a post-marketing clinical study.

   Note: This does not apply to participants participating in observational studies without interventional or surgical therapy.
2. The participant previously received therapy with azilsartan.
3. The participant has poorly controlled hypertension indicated by an office sitting systolic blood pressure higher by at least 22 mmHg and/or an office sitting diastolic blood pressure higher by at least 17 mmHg than the 95th percentiles of the reference blood pressure values of children by gender and age.
4. The participant has a diagnosis of malignant or accelerated hypertension.
5. The participant was noncompliant (compliance: <70% or >130%) with the study drug during the Run-in Period. The proportion of the number of the received the study drug to the number of the study drug which the participants should receive.
6. The participant has severe renal dysfunction (eGFR <30 mL/min/1.73 m^2), is receiving dialysis, has a renovascular disease affecting one or both kidneys, severe nephrotic syndrome not in remission, or a serum albumin level <2.5 g/dL.
7. The participant has a history of, or the signs/symptoms of serious cardiovascular, hepatobiliary, gastrointestinal, endocrine (eg, hyperthyroidism, Cushing's syndrome), hematological, immunological, urogenital, psychiatric disease, cancer, or any other disease that adversely affects participant's health, or, in the opinion of the investigator or subinvestigator, potentially confounds the study results.
8. The participant has hemodynamically significant left ventricular outflow obstruction due to aortic stenosis or uncorrected aortic valvular disease, or is scheduled to undergo a medical procedure affecting blood pressure during the study (eg, correction of arterial anomaly).

   Note: This does not apply to participants who received medical procedure(s) (eg, surgery for aortic coarctation) before the study and investigator or subinvestigator assess that participant's condition is stable at screening.
9. The participant has a history of or concurrent clinically significant abnormality of 12-lead ECG that, in the opinion of the investigator or subinvestigator, disqualifies the participant for participation in the study.
10. The participant has poorly controlled diabetes mellitus indicated by HbA1c >9.0% at screening.
11. The participant has an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level >=2.5 × the upper limit of normal (ULN), or a total bilirubin level >=1.5 × ULN at screening, severely impaired hepatic function, any active liver disease (regardless of the cause), or jaundice.
12. The participant has hyperkalemia exceeding ULN at screening.
13. The participant has a history of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection at screening.
14. The participant has a known hypersensitivity or allergy to any ARBs.
15. The participant needs treatment with any of the excluded medication.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (19):
- Japan (19):
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Aichi Children's Health and Medical Center, Ōbu, Aichi-ken
  - Hyogo Prefectural Kobe Children's Hospital, Kobe, Hyōgo
  - National Hospital Organization Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Miyagi Children's Hospital, Sendai, Miyagi
  - Tohoku University Hospital, Sendai, Miyagi
  - University of the Ryukyus Hospital, Nakagami-gun, Okinawa
  - Okinawa Prefectural Nanbu Medical Center & Children's Medical Center, Shimajiri-gun, Okinawa
  - Osaka University Hospital, Suita, Osaka
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Tokyo Metropolitan Hospital Organization Tokyo Metropolitan Children's Medical Center, Fuchū, Tokyo
  - National Center for Child Health and Development, Setagaya-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Hiroshima Prefectural Hospital, Hiroshima
  - Local Independent Administrative Institution Saitama prefectural hospital organization Saitama Children's Medical Center, Saitama
  - Shizuoka Childrens Hospital, Shizuoka
  - Wakayama Medical University Hospital, Wakayama

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5fd8c7110faaff002927fb7a

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 19 investigative sites in Japan from 17 May 2021 to 28 December 2023.
Pre-assignment Details: Participants with hypertension were enrolled in the study to receive TAK-536. The study consisted of a 2-week Run-in Period to receive placebo, followed by a 52-week Treatment Period to receive TAK-536, orally, once daily.
Groups:
- Run-in Period: Placebo: TAK-536 matching-placebo, orally, once daily, before or after breakfast for up to 2 weeks.
- Treatment Period: TAK-536 0.1 mg/kg - 0.8 mg/kg: TAK-536 0.1 milligram per kilogram (mg/kg) (not exceeding 2.5 milligram per day [mg/day]), granules, orally, once daily, before or after breakfast on Day 1 for up to 52 weeks. The dose was titrated to the highest dose of 0.8 mg/kg (not exceeding 20 mg/day) as needed and based on body weight.
Period: Run-in Period (2 Weeks)
Arm/Group | Run-in Period: Placebo | Treatment Period: TAK-536 0.1 mg/kg - 0.8 mg/kg
Started | 10 | 0
Completed | 9 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Treatment Period (52 Weeks)
Arm/Group | Run-in Period: Placebo | Treatment Period: TAK-536 0.1 mg/kg - 0.8 mg/kg
Started | 0 | 9 (The participants whose blood pressure meet the inclusion and exclusion criteria after receiving placebo in the Run-in Period entered the Treatment Period to receive TAK-536.)
Completed | 0 | 7
Not Completed | 0 | 2
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received the placebo in the Run-in Period.
Arm/Group | Run-in Period: Placebo
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 10
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced At Least One Treatment-Emergent Adverse Event (TEAE)
Description: An Adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant whose parent or legal guardian had signed informed consent form to participate in a study; it did not necessarily have to have a causal relationship with this treatment or study participation. An AE could therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the study participation whether or not it was considered related to the drug or study procedures. A TEAE was defined as any AE occurring after the start of TAK-536 administration, and until the end of follow-up period of 2 weeks.
Time Frame: From first dose of study drug up to end of follow-up period (Week 54)
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of study drug for the Treatment Period. As per planned analysis, outcomes in this study were analysed, collected and reported for treatment period only.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: TAK-536 0.1 mg/kg - 0.8 mg/kg
Number analyzed (Participants) | 9
Participants | 9

2. Primary Outcome: Number of Participants With TEAE Related to Resting 12-lead Electrocardiogram (ECG)
Description: The relatedness of TEAEs with resting 12-lead ECG was based upon investigator discretion.
Time Frame: From first dose of study drug up to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: TAK-536 0.1 mg/kg - 0.8 mg/kg
Number analyzed (Participants) | 9
Participants | 0

3. Primary Outcome: Number of Participants With TEAE Related to Anthropometric Measurement
Description: The anthropometric measurements included weight, height and body mass index (BMI). The relatedness of TEAEs to anthropometric measurements was based upon investigator discretion.
Time Frame: From first dose of study drug up to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: TAK-536 0.1 mg/kg - 0.8 mg/kg
Number analyzed (Participants) | 9
Participants | 0

4. Primary Outcome: Number of Participants With TEAE Related to Clinical Laboratory Parameters
Description: The laboratory values outside the range (triglycerides greater than [>] 2.5*upper limit of normal [ULN], blood urea nitrogen [BUN] >30 milligram per deciliter [mg/dL], estimated glomerular filtration rate [eGFR] less than [<] 30 milliliter per minute per 1.73 square meter [mL/min/1.73m^2], and glucose <50 mg/dL were considered markedly abnormal for TEAEs. The relatedness of TEAEs to clinical laboratory parameters was based upon investigator discretion.
Time Frame: From first dose of study drug up to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: TAK-536 0.1 mg/kg - 0.8 mg/kg
Number analyzed (Participants) | 9
Participants | 3

5. Primary Outcome: Number of Participants With TEAE Related to Vital Sign Values
Description: Vital signs included home sitting blood pressure (diastolic and systolic) and office sitting pulse rate (pulse rate per 1 minute). The pulse rate measured at the last measurement of the sitting blood pressure was used as the sitting pulse rate value. The relatedness of TEAEs to vital signs was based upon investigator discretion.
Time Frame: From first dose of study drug up to end of follow-up period (Week 54)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: TAK-536 0.1 mg/kg - 0.8 mg/kg
Number analyzed (Participants) | 9
Participants | 1

6. Secondary Outcome: Change From Baseline in Office Trough Sitting Diastolic Blood Pressure at Weeks 12 (Last Observation Carried Forward [LOCF]) and 52 (LOCF)
Description: Office trough sitting diastolic blood pressure were measured in a sitting position. LOCF method was used to impute missing values.
Time Frame: Baseline, Weeks 12 (LOCF) and 52 (LOCF)
Population: The full analysis set (FAS) included all participants who were enrolled and received at least 1 dose of study drug for the Treatment Period. As per planned analysis, outcomes in this study were analysed, collected and reported for treatment period only.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Treatment Period: TAK-536 0.1 mg/kg - 0.8 mg/kg
Number analyzed (Participants) | 9
millimeters of mercury (mmHg)
  Change from Baseline at Week 12 (LOCF) | -10.9 (11.04)
  Change from Baseline at Week 52 (LOCF) | -14.8 (8.39)

7. Secondary Outcome: Change From Baseline in Office Trough Sitting Systolic Blood Pressure at Weeks 12 (LOCF) and 52 (LOCF)
Description: Office trough sitting systolic blood pressure were measured in a sitting position. LOCF method was used to impute missing values.
Time Frame: Baseline, Weeks 12 (LOCF) and 52 (LOCF)
Population: The FAS included all participants who were enrolled and received at least 1 dose of study drug for the Treatment Period. As per planned analysis, outcomes in this study were analysed, collected and reported for treatment period only.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Period: TAK-536 0.1 mg/kg - 0.8 mg/kg
Number analyzed (Participants) | 9
mmHg
  Change from Baseline at Week 12 (LOCF) | -8.0 (6.73)
  Change from Baseline at Week 52 (LOCF) | -10.9 (8.30)

8. Secondary Outcome: Percentage of Participants Who Achieved the Target Blood Pressure at Weeks 12 (LOCF) and 52 (LOCF)
Description: The target blood pressure was defined as the normal reference range for blood pressure by age according to guidelines on the clinical examination for decision making of diagnosis and drug therapy in pediatric participants with cardiovascular diseases by the Japanese Circulation Society 2018 (JCS 2018). LOCF method was used to impute missing values.
Time Frame: At Weeks 12 (LOCF) and 52 (LOCF)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Period: TAK-536 0.1 mg/kg - 0.8 mg/kg
Number analyzed (Participants) | 9
percentage of participants
  At Week 12 (LOCF) | 44.4 [13.700 to 78.799]
  At Week 52 (LOCF) | 44.4 [13.700 to 78.799]

9. Secondary Outcome: Plasma Concentration of TAK-536
Description: Plasma concentration of TAK-536 were reported.
Time Frame: Weeks 2, 4, 8 and 12: Pre-dose and at 2 hours post-dose; Week 16: 2 hours post-dose
Population: The FAS included all participants who were enrolled and received at least 1 dose of study drug for the Treatment Period. Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure and 'number of participants analyzed' refer to the participants evaluable for specified time points. As per planned analysis, outcomes in this study were analysed, collected and reported for treatment period only.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Treatment Period: TAK-536 0.1 mg/kg - 0.8 mg/kg
Number analyzed (Participants) | 8
nanogram per milliliter (ng/mL)
  At Week 2 (Pre-dose): number analyzed (Participants) | 5
  At Week 2 (Pre-dose) | 14.0 (11.96)
  At Week 2 (Post-dose): number analyzed (Participants) | 2
  At Week 2 (Post-dose) | 356.0 (435.58)
  At Week 4 (Pre-dose): number analyzed (Participants) | 4
  At Week 4 (Pre-dose) | 42.5 (25.77)
  At Week 4 (Post-dose): number analyzed (Participants) | 1
  At Week 4 (Post-dose) | 728.0 (NA) — Standard deviation could not be calculated for 1 participant.
  At Week 8 (Pre-dose): number analyzed (Participants) | 2
  At Week 8 (Pre-dose) | 50.0 (8.49)
  At Week 8 (Post-dose): number analyzed (Participants) | 0
  At Week 12 (Pre-dose): number analyzed (Participants) | 1
  At Week 12 (Pre-dose) | 170.0 (NA) — Standard deviation could not be calculated for 1 participant.
  At Week 12 (Post-dose): number analyzed (Participants) | 0
  At Week 16 (Post-dose) | 2374.5 (1924.50)

ADVERSE EVENTS:
Time Frame: Run-in Period: From first dose in Run-in Period up to 2 weeks; Treatment Period: From first dose in Treatment Period up to end of follow-up period (54 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. AEs were not collected by dose level. As planned, combined dose-wise data of all TAK-536 doses (0.1 mg/kg - 0.8 mg/kg) was collected, analyzed and reported for Treatment Period.
Groups:
- TAK-536 0.1 mg/kg - 0.8 mg/kg: TAK-536 0.1 mg/kg (not exceeding 2.5 mg/day), granules, orally, once daily, before or after breakfast on Day 1 for up to 52 weeks in Treatment Period. The dose was titrated to the highest dose of 0.8 mg/kg (not exceeding 20 mg/day) as needed and based on body weight.
Arm/Group | Run-in Period: Placebo | TAK-536 0.1 mg/kg - 0.8 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 4/9
Other Adverse Events (participants affected / at risk) | 3/10 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Period: Placebo (N=10) | TAK-536 0.1 mg/kg - 0.8 mg/kg (N=9)
Acute kidney injury (Renal and urinary disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 1
Coronavirus infection (Infections and infestations) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Period: Placebo (N=10) | TAK-536 0.1 mg/kg - 0.8 mg/kg (N=9)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
BK virus infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Hangnail (Skin and subcutaneous tissue disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Impetigo (Infections and infestations) | 0 | 1
Infected aural fistula (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 7
Pollakiuria (Renal and urinary disorders) | 0 | 1
Pruritus genital (Reproductive system and breast disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT04668157/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/57/NCT04668157/SAP_001.pdf